CLINICAL TRIAL: NCT05365451
Title: Pharmacokinetic Drug-Drug Interaction Study to Identify Biomarkers of Kidney Transporters
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Mary Paine, Professor, Washington State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19163; R01HD081299 (NIH)
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Interaction; Endogenous Biomarkers
Keywords: Kidney Transporter; Pharmacokinetics
MeSH Terms: interventions — Metformin; Cimetidine; Furosemide; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1A: metformin alone (baseline) (Experimental): Arm 1A will consist of administration of a single dose of metformin (50 mg) by mouth as a liquid to 16 subjects (8 males, 8 females). Plasma and urine will be collected from 0-24 hours. Participants may or may not elect to participate in Arms 2A and 2B. A washout of at least 7 days will occur between Arm 1A and Arm 1B.
  Interventions: Drug: MetFORMIN Oral Solution
- Arm 1B: metformin + cimetidine (Experimental): Arm 1B will consist of administration of a single oral dose of cimetidine (400 mg) with water by mouth. One hour later, metformin (50 mg) will be administered by mouth as a liquid. Plasma and urine will be collected from 0-24 hours. Participants may or may not elect to participate in Arms 2A and 2B. A washout of at least 7 days will occur between Arm 1B and Arm 2A.
  Interventions: Drug: MetFORMIN Oral Solution; Drug: Cimetidine 400 MG
- Arm 2A: furosemide alone (baseline) (Experimental): Arm 2A will consist of administration of a single dose of furosemide (5 mg) by mouth as a liquid. Plasma and urine will be collected from 0-24 hours. A washout of at least 7 days will occur between Arm 2A and Arm 2B.
  Interventions: Drug: Furosemide Oral Liquid Product
- Arm 2B: furosemide + probenecid (Experimental): Arm 2B will consist of administration of a single oral dose of probenecid (1,000 mg) with water by mouth. One hour later, furosemide (5 mg) will be administered by mouth as a liquid. Plasma and urine will be collected from 0-24 hours. Participants may or may not elect to participate in Arms 1A and 1B. A washout of at least 7 days will occur between Arm 2B and Arm 1A.
  Interventions: Drug: Furosemide Oral Liquid Product; Drug: Probenecid 500 MG

INTERVENTIONS:
Drug: MetFORMIN Oral Solution — liquid
  Other Names: Riomet
  Arms: Arm 1A: metformin alone (baseline); Arm 1B: metformin + cimetidine
Drug: Cimetidine 400 MG — tablet
  Other Names: Tagamet
  Arms: Arm 1B: metformin + cimetidine
Drug: Furosemide Oral Liquid Product — oral solution
  Other Names: Lasix
  Arms: Arm 2A: furosemide alone (baseline); Arm 2B: furosemide + probenecid
Drug: Probenecid 500 MG — tablet
  Other Names: Probalan
  Arms: Arm 2B: furosemide + probenecid

SUMMARY:
The objective of this study is to confirm the feasibility of using a panel of endogenous substrates/metabolites as a robust biomarker of OCTs and OATs by conducting a controlled, comprehensive clinical drug-drug interaction study in healthy adult volunteers. Metformin and furosemide will be used as probe drugs for OCTs and OATs, respectively; cimetidine and probenecid will be used as corresponding inhibitors. Results from this study will validate this novel approach, which will be extended to children by collaborators at Children's Mercy Hospital in Kansas City, MO.

DETAILED DESCRIPTION:
The kidneys are major organs responsible for the excretion of both endogenous and exogenous compounds, the latter including drugs and other xenobiotics. Excretion occurs via passive or active processes, the latter involving transporters such as organic cation transporters (OCTs) and organic anion transporters (OATs). Inhibition of these transporters, coupled with the large interindividual variability in transporter expression, can lead to toxic accumulation of compounds/xenobiotics cleared primarily by this route. During drug discovery and development, if in vitro evidence suggests renal transporters mediate excretion of a new chemical entity, the Food and Drug Administration recommends conducting a controlled clinical study to evaluate potential risks. These time-consuming and expensive clinical studies routinely involve adult participants and known substrates of renal transporters. However, such studies are not always feasible in children due to the enhanced potential for toxicities. This limitation led to the hypothesis that endogenous substrates could be used as surrogates, or biomarkers, of individual renal transporter function.

Endogenous OCT substrates, such as 1-methyladenosine (m1A) and 1-methylnicotinamide (MNA), as well as OATs, such as homovanillic acid (HVA) and pyridoxic acid (PDA), are promising biomarkers of renal transporters in adults. However, using one or few such endogenous substrates can be misleading due to factors other than variability in specific renal transporter function. We propose to address this knowledge gap by using a panel of endogenous substrates/metabolites that recently has been identified as a robust biomarker of rodent Octs and Oats. Validation of these substrates/metabolites as biomarkers of OCTs and OATs in humans, both adults and children, will aid in the development of physiologically-based pharmacokinetic models that can be used to predict renal transporter-mediated xenobiotic excretion, drug-drug interactions, and toxicity in children.

ELIGIBILITY:
Inclusion Criteria:

Are from 18-65 years old and healthy

* Are not taking any medications (prescription and non-prescription) or dietary/herbal supplements that can interfere with your ability to eliminate the study drugs from your body
* Are willing to stop taking dietary/herbal supplements and citrus juices for several weeks
* Are willing to stop consuming caffeinated beverages or other caffeine-containing products the evening before and the morning of the first day of each study arm
* Are willing to stop drinking alcoholic beverages for at least 1 day prior to any study day and during the study day
* Are willing to use an acceptable method of birth control that does not include oral contraceptive pills or patches (such as abstinence, copper IUD, condom) throughout your participation in the study and for at least 3 weeks after you last take the study drugs
* Have the time to participate

Exclusion Criteria:

* Are under 18 or over 65 years old
* Smoke/vape/chew tobacco products
* Use cannabis products, including marijuana, hemp, and other THC- and CBDcontaining products• Are taking medications or dietary/herbal supplements that can interfere with your ability to eliminate the study drugs from your body
* Have a chronic illness such as (but not limited to) kidney disease, liver disease, diabetes mellitus, high blood pressure, coronary artery disease, chronic obstructive pulmonary disease, cancer, or HIV/AIDS
* Have a hematologic (blood) disorder
* Have a history of drug or alcohol addiction or major psychiatric illness
* Have a history of allergy to metformin, cimetidine, furosemide, or probenecid
* Are pregnant, nursing, or plan to become pregnant within 3 weeks after participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University College of Pharmacy and Pharmaceutical Sciences, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morrissey KM, Stocker SL, Wittwer MB, Xu L, Giacomini KM. Renal transporters in drug development. Annu Rev Pharmacol Toxicol. 2013;53:503-29. doi: 10.1146/annurev-pharmtox-011112-140317. Epub 2012 Nov 8. PMID 23140242
- [Background] US Food and Drug Administration. Clinical Drug Interaction Studies - Cytochrome P450 Enzyme- and Transporter-Mediated Drug Interactions Guidance for Industry. https://www.fda.gov/regulatory-information/search-fda-guidance-documents/clinical-drug-interaction-studies-cytochrome-p450-enzyme-and-transporter-mediated-drug-interactions.
- [Background] Shen H, Holenarsipur VK, Mariappan TT, Drexler DM, Cantone JL, Rajanna P, Singh Gautam S, Zhang Y, Gan J, Shipkova PA, Marathe P, Humphreys WG. Evidence for the Validity of Pyridoxic Acid (PDA) as a Plasma-Based Endogenous Probe for OAT1 and OAT3 Function in Healthy Subjects. J Pharmacol Exp Ther. 2019 Jan;368(1):136-145. doi: 10.1124/jpet.118.252643. Epub 2018 Oct 25. PMID 30361237
- [Background] Miyake T, Mizuno T, Takehara I, Mochizuki T, Kimura M, Matsuki S, Irie S, Watanabe N, Kato Y, Ieiri I, Maeda K, Ando O, Kusuhara H. Elucidation of N 1-methyladenosine as a Potential Surrogate Biomarker for Drug Interaction Studies Involving Renal Organic Cation Transporters. Drug Metab Dispos. 2019 Nov;47(11):1270-1280. doi: 10.1124/dmd.119.087262. Epub 2019 Sep 11. PMID 31511257
- [Background] Naji-Talakar S, Sharma S, Martin LA, Barnhart D, Prasad B. Potential implications of DMET ontogeny on the disposition of commonly prescribed drugs in neonatal and pediatric intensive care units. Expert Opin Drug Metab Toxicol. 2021 Mar;17(3):273-289. doi: 10.1080/17425255.2021.1858051. Epub 2021 Jan 20. PMID 33256492
- [Background] Feng B, Varma MV. Evaluation and Quantitative Prediction of Renal Transporter-Mediated Drug-Drug Interactions. J Clin Pharmacol. 2016 Jul;56 Suppl 7:S110-21. doi: 10.1002/jcph.702. PMID 27385169

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin Alone, Then Cimetidine + Metformin, Then Furosemide Alone, Then Probenecid + Furosemide: 16 subjects were administered 50 mg metformin as a solution for Part 1 Arm A. The same 16 subjects were administered 400 mg cimetidine as a tablet, then 50 mg metformin as a solution for Part 1 Arm B. The same 16 subjects were administered 5 mg furosemide as a tablet for Part 2 Arm A. The same 16 subjects were administered 1000 mg probenecid as a tablet, then 5 mg furosemide as a tablet for Part 2 Arm B.
Period: Overall Study
Arm/Group | Metformin Alone, Then Cimetidine + Metformin, Then Furosemide Alone, Then Probenecid + Furosemide
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1A - Arm 2A - Arm 1B - Arm 2B: 16 subjects completed Part 1, Arms A and B, then Part 2, Arms A and B, in that order.
Arm/Group | Arm 1A - Arm 2A - Arm 1B - Arm 2B
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12
  Asian | 2
  Black | 1
  More than one race | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Metformin Area Under the Concentration vs. Time Curve (AUC)
Description: baseline metformin area under the concentration vs. time curve (AUC)
Time Frame: 0-24 hours
Measure: Geometric Mean (90% Confidence Interval); unit: mcg*h/L
Arm/Group | Arm 1A - Arm 2A - Arm 1B - Arm 2B
Number analyzed (Participants) | 16
mcg*h/L | 830 [710 to 970]

2. Primary Outcome: Metformin AUC in Presence of Cimetidine
Description: Metformin area under the concentration vs. time curve (AUC) in presence of cimetidine
Time Frame: 0-24 hours
Measure: Geometric Mean (90% Confidence Interval); unit: mcg*h/L
Arm/Group | Arm 1A - Arm 2A - Arm 1B - Arm 2B
Number analyzed (Participants) | 16
mcg*h/L | 1030 [875 to 1210]

3. Primary Outcome: Metformin Maximum Concentration (Cmax)
Description: baseline metformin maximum concentration (Cmax)
Time Frame: 0-24 hours
Measure: Geometric Mean (90% Confidence Interval); unit: mcg/L
Arm/Group | Arm 1A - Arm 2A - Arm 1B - Arm 2B
Number analyzed (Participants) | 16
mcg/L | 124 [107 to 143]

4. Primary Outcome: Metformin Cmax in Presence of Cimetidine
Description: metformin Cmax in the presence of cimetidine
Time Frame: 0-24 hours
Measure: Geometric Mean (90% Confidence Interval); unit: mcg/L
Arm/Group | Arm 1A - Arm 2A - Arm 1B - Arm 2B
Number analyzed (Participants) | 16
mcg/L | 168 [145 to 195]

5. Primary Outcome: Metformin Renal Clearance (CLr)
Description: baseline metformin renal clearance (CLr)
Time Frame: 0-24 hours
Measure: Geometric Mean (90% Confidence Interval); unit: L/h
Arm/Group | Arm 1A - Arm 2A - Arm 1B - Arm 2B
Number analyzed (Participants) | 16
L/h | 31 [27 to 34]

6. Primary Outcome: Metformin CLr in Presence of Cimetidine
Description: metformin CLr in the presence of cimetidine
Time Frame: 0-24 hours
Measure: Geometric Mean (90% Confidence Interval); unit: L/h
Arm/Group | Arm 1A - Arm 2A - Arm 1B - Arm 2B
Number analyzed (Participants) | 16
L/h | 28 [25 to 31]

7. Primary Outcome: Furosemide Area Under the Concentration vs. Time Curve (AUC)
Description: baseline furosemide area under the concentration vs. time curve (AUC)
Time Frame: 0-24 hours
Measure: Geometric Mean (90% Confidence Interval); unit: ng.h/mL
Arm/Group | Arm 1A - Arm 2A - Arm 1B - Arm 2B
Number analyzed (Participants) | 16
ng.h/mL | 462.4 [338.3 to 586.5]

8. Primary Outcome: Furosemide AUC in Presence of Probenecid
Description: furosemide AUC in the presence of probenecid
Time Frame: 0-24 hours
Measure: Geometric Mean (90% Confidence Interval); unit: ng.h/mL
Arm/Group | Arm 1A - Arm 2A - Arm 1B - Arm 2B
Number analyzed (Participants) | 16
ng.h/mL | 854.6 [608.5 to 1100.7]

9. Primary Outcome: Furosemide Renal Clearance (CLr)
Description: baseline furosemide renal clearance (CLr)
Time Frame: 0-24 hours
Measure: Geometric Mean (90% Confidence Interval); unit: mL/min
Arm/Group | Arm 1A - Arm 2A - Arm 1B - Arm 2B
Number analyzed (Participants) | 16
mL/min | 96.1 [68.7 to 123.5]

10. Primary Outcome: Furosemide CLr in Presence of Probenecid
Description: furosemide CLr in the presence of probenecid
Time Frame: 0-24 hours
Measure: Geometric Mean (90% Confidence Interval); unit: mL/min
Arm/Group | Arm 1A - Arm 2A - Arm 1B - Arm 2B
Number analyzed (Participants) | 16
mL/min | 33.4 [24.2 to 42.6]

ADVERSE EVENTS:
Time Frame: 10 months
Groups:
- Metformin Alone: 16 subjects were administered 50 mg metformin as a solution for Part 1 Arm A.
- Cimetidine + Metformin: The same 16 subjects were administered 400 mg cimetidine as a tablet, then 50 mg metformin as a solution for Part 1 Arm B.
- Furosemide Alone: The same 16 subjects were administered 5 mg furosemide as a tablet for Part 2 Arm A.
- Probenecid + Furosemide: The same 16 subjects were administered 1000 mg probenecid as a tablet, then 5 mg furosemide as a tablet for Part 2 Arm B.
Arm/Group | Metformin Alone | Cimetidine + Metformin | Furosemide Alone | Probenecid + Furosemide
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 1/16 | 3/16 | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin Alone (N=16) | Cimetidine + Metformin (N=16) | Furosemide Alone (N=16) | Probenecid + Furosemide (N=16)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
nausea/vomiting (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IV site tenderness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT05365451/Prot_SAP_000.pdf